CLINICAL TRIAL: NCT06008886
Title: Effect of a Vegan Diet Versus a Mediterrean Diet on Performance, Cardiorespiratory Fitness, Metabolic Health, Immune Status, and Environmental Impact in Healthy Adults
Brief Title: Effect of a Vegan Diet Versus a Mediterranean Diet. Assessing Health Outcomes
Acronym: OMNIVEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, Miguel López Moreno, Principal Investigator, Universidad Francisco de Vitoria
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20/2023
Record Dates: First submitted 2023-07-28; First posted 2023-08-24 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-08

CONDITIONS: Cardiometabolic Syndrome
Keywords: Plant-Based Diet; Environmental Impact; Cardiorespiratory Fitness; Performance; Metabolic Health; Mediterranean diet; Vegan diet
MeSH Terms: conditions — Metabolic Syndrome | interventions — Diet, Vegan; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegan diet (Experimental): Vegan diet all foods included were of plant sources. During the vegan diet, the participants took 1000 µg of cyanocobalamin twice a week (Harrison Sport Nutrition, Granada, Spain)
  Interventions: Behavioral: Vegan diet
- Mediterranean diet (Active Comparator): In the case of the mediterranean diet, foods of animal sources were also included (animal protein accounted for 60% of total protein intake). In this diet there was a predominance of plant foods; moderate to low consumption of fish, white meat, low-fat dairy and eggs; and very low consumption of red and processed meats, butter, full-fat dairy and sweets.
  Interventions: Behavioral: Mediterranean diet

INTERVENTIONS:
Behavioral: Vegan diet — Normocaloric diet based solely on foods of plant sources.
  Arms: Vegan diet
Behavioral: Mediterranean diet — Diet with a predominance of plant foods fruits, vegetables, whole grains, nuts and legumes); moderate to low consumption of fish, white meat, low-fat dairy and eggs; and very low consumption of red and processed meats, butter, full-fat dairy and sweets.
  Arms: Mediterranean diet

SUMMARY:
This study aimed to evaluate the effect of a vegan diet (supplemented with vitamin B12) and an mediterranean diet on performance, cardiorespiratory fitness, metabolic health, immune status, and environmental impact in healthy adults.

DETAILED DESCRIPTION:
OMNIVEG is a controlled crossover trial. Initially, registered dietitians conducted an assessment of participants' lifestyles in a preliminary session. Qualified nutritionists then developed personalized diets for each participant in accordance with the recommendations of the International Society of Sports Nutrition (ISSN). These diets followed specific guidelines, including a daily intake of 3-5 g of carbohydrates per kilogram of body weight, 1.4-2.0 g of protein per kilogram of body weight, and 0.5-1.5 g of fat per kilogram of body weight.

Both the mediterranean diet and vegan diets prescribed to the participants were isocaloric, with similar distributions of macronutrients. The primary difference between the two interventions was the source of food: the vegan diet exclusively comprised plant-based foods, while the omnivorous diet included foods of both animal and plant sources. In the case of the omnivorous diet, 60% of the total protein intake was derived from animal sources (mainly from fish, white meat, low-fat dairy and eggs).

As part of the vegan diet, participants were instructed to take 1000 µg of cyanocobalamin (a form of vitamin B12) twice a week from Harrison Sport Nutrition, Granada, Spain. This supplementation aimed to ensure adequate vitamin B12 intake, which is essential for individuals following a vegan diet.

Throughout the study period, participants were advised to maintain their initial physical exercise frequency and volume to maintain consistency and avoid confounding variables. To ensure standardized measurements, all tests were conducted in the same laboratory, employing identical testing devices, and supervised by the same group of researchers. This approach aimed to minimize experimental variability and improve the reliability of the study's results.

ELIGIBILITY:
Inclusion Criteria:

* Men.
* Aged between 18-40 years.
* Physically active according to the recommendations of the World Health Organization (WHO).
* Body Mass Index (BMI) between 18.5-24.9 kg/m2.
* No tobacco use.
* No or low alcohol consumption and no orthopedic limitations that would interfere with the performance of the study tests.

Exclusion Criteria:

* Chronic diseases that impair athletic performance (cardiovascular, metabolic, gastrointestinal, respiratory) within the last six months.
* Musculoskeletal disease within the last six months.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | 4 weeks
  Cardiorespiratory fitness was measured using Maximal oxygen uptake (VO2max).
Metabolic health | 4 weeks
  Metabolic health was measured using serum total cholesterol (TC), cholesterol-LDL (LDL-c) and colesterol-HDL (HDL-c)
Performance | 4 weeks
  Performance was measured using FATmax (g/min).
Performance | 4 weeks
  Performance was measured using countermovement (CMJ) (W) and squat jump (SJ).
Performance | 4 weeks
  Performance was measured using squat jump (SJ) (W)
Environmental impact assessment | 4 weeks
  Environmental impact was measured using Global-warming potential-100
Inmune status | 4 weeks
  Inmune status was measured using lymphocyte levels (109/L )

SECONDARY OUTCOMES:
Performance | 4 weeks
  Performance was measured using handgrip
Metabolic health | 4 weeks
  Metabolic health was measured using systolic blood pressure (SBP) and diastolic blood pressure (DBP).
Inmune status | 4 weeks
  Inmune status was measured using monocyte, eosinophils and neutrophils levels (10^9/L)
Environmental impact assessment | 4 weeks
  Environmental impact was measured using blue water footprint and land use.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel López Moreno, Phd, Principal Investigator — Universidad Francisco de Vitoria
Locations (1):
- Francisco de Vitoria University, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Moreno M, Fresan U, Del Coso J, Munoz A, Aguilar-Navarro M, Iglesias-Lopez MT, Amaro-Gahete FJ, Gutierrez-Hellin J. The OMNIVEG Study: Effects of Transitioning from a Traditional to a Vegan Mediterranean Diet on Fat Oxidation During Exercise. Nutrients. 2025 Jul 9;17(14):2274. doi: 10.3390/nu17142274. PMID 40732902
- [Derived] Lopez-Moreno M, Fresan U, Del Coso J, Aguilar-Navarro M, Iglesias Lopez MT, Pena-Fernandez J, Munoz A, Gutierrez-Hellin J. The OMNIVEG STUDY: Health outcomes of shifting from a traditional to a vegan Mediterranean diet in healthy men. A controlled crossover trial. Nutr Metab Cardiovasc Dis. 2024 Dec;34(12):2680-2689. doi: 10.1016/j.numecd.2024.08.008. Epub 2024 Aug 23. PMID 39358106